CLINICAL TRIAL: NCT06423001
Title: A Randomized, Cross-over, Placebo-Controlled, Double-Blind Clinical Trial on the Efficacy and Safety of Oral Administration of Postibiotic by FOS Fermentation From Lactobacillus Paracasei in the Treatment of Irritable Bowel Syndrome.
Brief Title: Efficacy and Safety of Oral Administration of Postibiotic by FOS Fermentation From Lactobacillus Paracasei in the Treatment of Irritable Bowel Syndrome.
Acronym: prePO23
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: ID 2939
Record Dates: First submitted 2024-04-24; First posted 2024-05-21 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-04

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PostbiotiX Slowing (Treatment A) Sequence AB (Experimental): Each patient will be supplied with the investigational product at Visit 0 (V0, Kit V0, PostibiotiX Slowing) and at visit 3 (V3, Kit V3, Placebo), based on the outcome of the randomization at V0 (Sequence AB, PostbiotiX Slowing/Placebo).
  Interventions: Dietary Supplement: PostbiotiX Slowing 4 g sachets PostbiotiX Slowing is a food supplement based on Fermented FOS from Lactobacillus paracasei CNCM I-5220.
- Placebo (Tratment B) Sequence BA (Experimental): Each patient will be supplied with the investigational product at Visit 0 (V0, Kit V0, Placebo) and at visit 3 (V3, Kit V3, PostibiotiX Slowing), based on the outcome of the randomization at V0 (Sequence BA, Placebo/PostbiotiX Slowing).
  Interventions: Dietary Supplement: PostbiotiX Slowing 4 g sachets PostbiotiX Slowing is a food supplement based on Fermented FOS from Lactobacillus paracasei CNCM I-5220.

INTERVENTIONS:
Dietary Supplement: PostbiotiX Slowing 4 g sachets PostbiotiX Slowing is a food supplement based on Fermented FOS from Lactobacillus paracasei CNCM I-5220. — Each patient will be supplied with the investigational product at Visit 0, PostibiotiX Slowing and at visit 3, based on the outcome of the randomization at V0 (Sequence AB, PostbiotiX Slowing/Placebo; Sequence BA, Placebo/PostbiotiX Slowing).

SUMMARY:
Irritable bowel syndrome (IBS) is a highly prevalent functional pathology which currently has no real standardized and effective therapy, despite having a significant impact on quality of life and on social-health costs.

Post-biotics have demonstrated in various in vitro and in vivo studies the ability to modulate the microbiota, the intestinal barrier function, the immune response as well as having systemic effects, with prospects for good efficacy in treatment of IBS.

DETAILED DESCRIPTION:
PostbiotiX Slowing is a food supplement based on Fermented FOS from Lactobacillus paracasei CNCM I-5220, mallow and chamomile.

The Fermented FOS from Lactobacillus paracasei CNCM I-5220 (postbiotic) is the result of a controlled fermentation. The fermentation process allows to eliminate all the individual variability that depends on the microbiota, the diet and the psycho-physical conditions of the single individual, offering a mixture of bacterial metabolites and fermented fiber (postbiotic), which has the functional activity. In addition, as FOS is already fermented it does not induce the formation of gas typical of fiber fermentation in IBS patients, thus providing all the beneficial effects of the fiber without its side effects.

The fermented FOS from Lactobacillus paracasei CNCM I-5220 (postbiotic) is easily absorbed by the gut.

Dosage and method of use: PostbiotiX Slowing 4 g sachets, administered at the dosage of one sachet a day. To pour the contents of the sachet in a glass, add 150 ml of water, mix until complete dissolution of the powder and taken immediately, preferably as soon as awakened, and away from meals.

Ingredients: Maltodextrin, Aroma, Fermented FOS from Lactobacillus paracasei CNCM I-5220, mallow (Malva sylvestris L.) flowers and leaves d.e. tit. 20% polysaccharides, chamomile (Matricaria chamomilla L.) flowers d.e. tit. 0.3% apigenin, acidity regulator: citric acid; anti-caking agent: silicon dioxide; sweetener: sucralose.

Conservation method: to be kept in a cool and dry place, away from light, humidity, and direct sources of heat.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* IBS diagnosis according to ROME IV criteria
* Mild-moderate disease defined by IBS-SSS questionnaire at the baseline visit and after the washout period
* Signed Informed Consent
* Patients' ability to comply with the study procedures
* Stable diet within two months prior to the screening visit
* Negative colonoscopy (only > 50 years old patients)

Exclusion Criteria:

* Therapy with drugs or supplements included in the prohibited list
* Malignancy or history of malignancy, except patients with a history of surgically removed extraintestinal malignancy and a 5-year disease-free interval
* Unstable psychiatric pathology
* Organic bowel disease
* Major abdominal surgery, except appendectomy and cholecystectomy
* Relevant organic, systemic, metabolic pathologies or significant laboratory test abnormalities
* Pregnant or nursing women
* Patients with known hypersensitivity to one or more components of the product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in symptom intensity | 10 weeks
  Evaluated using a symptom measurement scale, at each visit, on a 4-point Likert scale (IBS symptom scale; 4 symptoms for a minimum sum score of 0, maximum 12).

SECONDARY OUTCOMES:
Change from baseline in IBS-SSS (symptom severity score) | up to 4 weeks
  IBS-SSS is a five-item questionnaire measuring frequency and intensity of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and the interference of IBS with daily life, scoring from 0 to 500.
Adequate overall symptom relief after treatment, | up to 10 days
  To assess adequate overall relief, patients will be asked weekly to answer the question "Compared to how you usually felt before taking the treatment, how would you rate your symptom relief (abdominal pain, bowel habits, and other symptoms of IBS) in the past 10 days?" Possible answers: 1, very relieved; 2, relieved; 3, somewhat relieved; 4, unchanged; 5, slightly worsened; 6, worsened; 7, much worsened.
Change from baseline after treatment in NRS: | up to 10 days
  Severity score of each of the individual symptoms included in the IBS-SSS (VAS sub-scores), assessed by numeric rating scale (NRS) from 0 to 100
Change from baseline after treatment in QqL: | up to 10 days
  Quality of life as assessed by IBS-QoL:
  The individual responses to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life
Change from baseline after treatment in HADS: | up to 10 days
  Hospital anxiety and depression scale (HADS):
  HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Fecal metagenomics: | up to 10 days
  Additional functional parameters in stool analysis differences before and after treatment (for example: digestive residues, bile acids, proteic composition)
Analyses of metabolomic: | up to 10 days
  Differences before and after treatment in the Sieric/plasma molecules such as for example Zonulin, soluble CD14, plasmatic inflammatory cytokines, bacterial DNA in the blood, and PBMCs analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lacy BE, Pimentel M, Brenner DM, Chey WD, Keefer LA, Long MD, Moshiree B. ACG Clinical Guideline: Management of Irritable Bowel Syndrome. Am J Gastroenterol. 2021 Jan 1;116(1):17-44. doi: 10.14309/ajg.0000000000001036. PMID 33315591
- [Background] Oka P, Parr H, Barberio B, Black CJ, Savarino EV, Ford AC. Global prevalence of irritable bowel syndrome according to Rome III or IV criteria: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2020 Oct;5(10):908-917. doi: 10.1016/S2468-1253(20)30217-X. Epub 2020 Jul 20. PMID 32702295
- [Background] Inadomi JM, Fennerty MB, Bjorkman D. Systematic review: the economic impact of irritable bowel syndrome. Aliment Pharmacol Ther. 2003 Oct 1;18(7):671-82. doi: 10.1046/j.1365-2036.2003.t01-1-01736.x. PMID 14510740
- [Background] Camilleri M. Management Options for Irritable Bowel Syndrome. Mayo Clin Proc. 2018 Dec;93(12):1858-1872. doi: 10.1016/j.mayocp.2018.04.032. PMID 30522596
- [Background] Salminen S, Collado MC, Endo A, Hill C, Lebeer S, Quigley EMM, Sanders ME, Shamir R, Swann JR, Szajewska H, Vinderola G. The International Scientific Association of Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of postbiotics. Nat Rev Gastroenterol Hepatol. 2021 Sep;18(9):649-667. doi: 10.1038/s41575-021-00440-6. Epub 2021 May 4. PMID 33948025
- [Background] Tsilingiri K, Barbosa T, Penna G, Caprioli F, Sonzogni A, Viale G, Rescigno M. Probiotic and postbiotic activity in health and disease: comparison on a novel polarised ex-vivo organ culture model. Gut. 2012 Jul;61(7):1007-15. doi: 10.1136/gutjnl-2011-300971. Epub 2012 Feb 1. PMID 22301383
- [Background] Tsilingiri K, Rescigno M. Postbiotics: what else? Benef Microbes. 2013 Mar 1;4(1):101-7. doi: 10.3920/BM2012.0046. PMID 23271068
- [Background] Aguilar-Toala JE, Arioli S, Behare P, Belzer C, Berni Canani R, Chatel JM, D'Auria E, de Freitas MQ, Elinav E, Esmerino EA, Garcia HS, da Cruz AG, Gonzalez-Cordova AF, Guglielmetti S, de Toledo Guimaraes J, Hernandez-Mendoza A, Langella P, Liceaga AM, Magnani M, Martin R, Mohamad Lal MT, Mora D, Moradi M, Morelli L, Mosca F, Nazzaro F, Pimentel TC, Ran C, Ranadheera CS, Rescigno M, Salas A, Sant'Ana AS, Sivieri K, Sokol H, Taverniti V, Vallejo-Cordoba B, Zelenka J, Zhou Z. Postbiotics - when simplification fails to clarify. Nat Rev Gastroenterol Hepatol. 2021 Nov;18(11):825-826. doi: 10.1038/s41575-021-00521-6. No abstract available. PMID 34556825
- [Background] Ma L, Tu H, Chen T. Postbiotics in Human Health: A Narrative Review. Nutrients. 2023 Jan 6;15(2):291. doi: 10.3390/nu15020291. PMID 36678162
- [Background] Adams CA. The probiotic paradox: live and dead cells are biological response modifiers. Nutr Res Rev. 2010 Jun;23(1):37-46. doi: 10.1017/S0954422410000090. Epub 2010 Apr 20. PMID 20403231